CLINICAL TRIAL: NCT05143853
Title: Does Additional Horizontal Fixation After Arthroscopically Assisted Coracoclavicular Stabilisation Matter in Final Outcome Measures: a Prospective Randomised Clinical Trial
Brief Title: HORizontal Instability AC Joint Study: A Prospective Randomised Clinical Trial
Acronym: HORAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Miha Ambrožič, Principal Investigator, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MAmbrozic
Record Dates: First submitted 2021-04-29; First posted 2021-12-03 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Acromioclavicular Separation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group with tape augmentation of acromioclavicular (AC) joint (Active Comparator): patients randomised in this group will have additional tape fixation around AC joint. Both groups will however have fixation in CC area.
  Interventions: Procedure: non-absorbable tape fixation around AC joint; Procedure: coracoclavicular (CC) fixation
- group without tape augmentation of AC joint (Sham Comparator): patients randomised in this group will not have additional tape fixation around AC joint. Both groups will however have fixation in CC area.
  Interventions: Procedure: no fixation around AC joint; Procedure: coracoclavicular (CC) fixation

INTERVENTIONS:
Procedure: non-absorbable tape fixation around AC joint — fixation around AC joint with tape in different configurations
  Arms: group with tape augmentation of acromioclavicular (AC) joint
Procedure: no fixation around AC joint — there will be no additional fixation around AC joint in this group
  Arms: group without tape augmentation of AC joint
Procedure: coracoclavicular (CC) fixation — mandatory coracoclavicular fixation with to suspensory systems, comprised of non-absorbable tapes and metal buttons

SUMMARY:
Comparing different treatement strategies in augmenting clavicle stabilisation

ELIGIBILITY:
Inclusion Criteria:

* consensus indication for surgical treatment of AC syndesmolysis
* OP in 3 weeks after injury
* patient age between 16 and 65 years
* normal shoulder function before injury

Exclusion Criteria:

* open injury
* ipsilateral arm/shoulder girdle/hand injuries
* very low patient's physical demands
* previous injuries of the affected area
* Rockwood classification 1, 2, or 6

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Constant-Murley score, minimum score 1, maximum score 100 (higher = better) | 1 year
  patient-reported outcome measure (PROM)

SECONDARY OUTCOMES:
SACS - specific AC score, minimum score 1, maximum score 100 (higher = better) | 1 year
  PROM
Horizontal RTG measurements, measured in mm | 1 year
  Overlap length (OL)
Horizontal RTG measurements, measured in mm2 | 1 year
  Overlap area (OA)

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided